CLINICAL TRIAL: NCT02293317
Title: A Phase II, Randomized, Placebo-Controlled, Double-Blind Study to Assess the Safety and Immunogenicity of Multimeric-001 Influenza Vaccine, Followed by a Seasonal Trivalent Influenza Vaccine (TIV)
Brief Title: Phase II Study to Assess Safety & Immunogenicity of Multimeric-001 Influenza Vaccine, Followed by TIV
Acronym: BVX006
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BiondVax Pharmaceuticals ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BVX-006
Record Dates: First submitted 2014-11-09; First posted 2014-11-18 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2014-11

CONDITIONS: Influenza
Keywords: Influenza Prime universal vaccine M-001 Multimeric
MeSH Terms: conditions — Influenza, Human | interventions — PN M001; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- M-001 0.5mg & TIV (Experimental): M-001 (0.5mg) administered intramuscular 3 times at 21 days intervals followed by vaccination with Trivalent Influenza Vaccine (TIV)
  Interventions: Biological: M-001; Drug: TIV
- M-001 1.0mg & TIV (Experimental): M-001 (1.0mg) administered intramuscular 3 times at 21 days intervals followed by vaccination with Trivalent Influenza Vaccine (TIV)
  Interventions: Biological: M-001; Drug: TIV
- Placebo & TIV (Placebo Comparator): 0.3ml Saline administered Intramuscular 3 times at 21 days intervals followed by vaccination with Trivalent Influenza Vaccine (TIV)
  Interventions: Drug: TIV; Other: Saline

INTERVENTIONS:
Biological: M-001 — A recombinant epitope based universal vaccine against seasonal and pandemic influenza
  Other Names: Multimeric-001
  Arms: M-001 0.5mg & TIV; M-001 1.0mg & TIV
Drug: TIV — HA based seasonal influenza vaccine, for 2014/15 seson
Other: Saline — Placebo
  Arms: Placebo & TIV

SUMMARY:
This is a single-site, randomized, double-blind, placebo-controlled study of Multimeric-001 in thirty six (36) volunteers 50-65 years of age.

All subjects will receive an intramuscular (IM) injection, in each one of three visits, with a 21±2 days interval between treatments.

DETAILED DESCRIPTION:
Subjects will undergo screening procedures within 30 days prior to first vaccination which will include medical history, vital signs, ECG, physical examination and safety blood and urine lab tests.

On the first treatment visit, eligible subjects will undergo pre-dose physical examination and vital signs, and a blood sample will be drawn for baseline cellular immunogenicity and circulating Interferon gamma (IFN-g). They will then receive an IM injection of either vaccine or placebo, according to the above treatment assignment, into the deltoid muscle preferably of the same arm. The subjects will remain under medical supervision for 2 hrs (± 15 min) at which time they will be released from the Clinical research center.

The second treatment will take place 21 (±2) days after the first vaccination. Procedures will be the same as that of Visit 2 Additional two follow-up visits will take place at approximately 24 hrs and 48h The third treatment will take place 21 (±2) days after the second vaccination. Procedures will be the same as that of Visit 2 21 days later, each subject will be immunized with the seasonal influenza vaccine approved for 2014/15 year.

A Study Termination visit will take place at 21 (±2) days after last vaccination. Adverse events (AEs) and changes in concomitant medications will be recorded, vital signs will be measured and the subjects will undergo physical examination and ECG. Blood and urine samples will be collected for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between ≥50 - ≤65 years old at the time expected for the first injection.
2. Eligible to receive the standard seasonal influenza vaccine according to the ministry of health guidelines.
3. Subjects who provide written informed consent to participate in the study.
4. Subjects able to adhere to the visit schedule and protocol requirements and are available to complete the study.
5. Pre-menopausal female subjects must have a negative serum pregnancy test at screening and be willing and able to use a medically acceptable method of birth control or declare that they are abstaining from sexual intercourse, from the screening visit through the study termination visit or be surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
6. Postmenopausal women, defined as women with menstruation cessation for 12 consecutive months prior to signing of the informed consent form.
7. Subjects must agree to use an acceptable contraceptive method the full term of the study period (including follow up).

Exclusion Criteria:

1. Subjects who are likely, in the opinion of the investigator, to confound the results of the study or may be exposed to additional risks by participation in the study, based on medical history, vital signs, ECG, physical examination and safety lab tests.
2. Subjects with known Guillain Barré Syndrome in the past.
3. Subjects who have been immunized with anti-influenza vaccine or infected by influenza virus (based on the assessment of the investigator) within eight months prior to first vaccination.
4. Known hypersensitivity associated with previous influenza vaccination.
5. Use of an influenza antiviral medication within 4 weeks of first vaccination.
6. Known allergy to egg protein
7. Known hypersensitivity and/or allergy to any drug or vaccine.
8. Persons deficient in producing antibodies, whether due to genetic defect, immunodeficiency disease, or immunosuppressive therapy.
9. History of any bleeding disorder or subjects with thrombocytopenia (since bleeding may occur following an intramuscular administration to these subjects).
10. Positive serology for Human immunodeficiency virus (HIV) , Hepatitis C Virus (HCV) antibody or HBsAg.
11. Any acute medical situation (e.g. acute infection, ongoing flu symptoms) with or without fever within 48 hours of vaccination, which is considered significant by the Investigator.
12. Pregnant or currently lactating women.
13. Subjects who participated in another interventional clinical study within 30 days prior to first dose.
14. Subjects who are non-cooperative or unwilling to sign consent form.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events in treatment vs control group | 3 months (from first visit to termination visit for each subject)
  Number of Participants with Adverse Events as a Measure of Safety and Tolerability will be measured in the experimental and control group, both local and systemic adverse events will be followed.

SECONDARY OUTCOMES:
Immunity induced by priming and boosting, measured by HAI (Hemagglutination Inhibition) | Day 84 (21 days after TIV injection)
  To characterize humoral immunity, Hemagglutination Inhibition (HAI) test for anti influenza antibodies to TIV strains will be measured after boosting with TIV, proportion of participants achieving seroconversion in the groups primed with M-001 and boosted with TIV, will be compared to participants given TIV alone.
Number of participants with cell mediated immune response in treatment vs control group | Day 63 (21 days after immunization with M-001)
  To characterize the cell mediated immune response, Fluorescence activated cell sorter (FACS) analysis for CD4/CD8 lymphocytes will be performed after 3 immunizations with M-001 as compared to the control group (injected 3 times with saline)

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Ben Yedidia, PhD, Study Chair — BiondVax Pharmaceuticals
Locations (1):
- Clinical Research Center, Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel